CLINICAL TRIAL: NCT07077590
Title: Can Labor Pain be Reduced by Open Placebo Intervention? A Bayesian Account for Labor Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roi Treister (Other)
Collaborators: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor-Investigator, Roi Treister, Prof. Roi Treister, PhD, University of Haifa
Organization: University of Haifa (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HINC-0091-24
Record Dates: First submitted 2025-05-07; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-05

CONDITIONS: Labor Pain and to Reduce Pain
Keywords: Labor pain; Open placebo; Within-subjects variability; personality
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (control arm) (No Intervention): Any woman who arrive to the labor room is connected to fluids (Hartman's solution), as part of routine care. In the control arm, the information given will be:" These fluids are important to keep your fluids balance, and is given to any delivering woman".
- Open placebo (Active Comparator): Any woman who arrive to the labor room is connected to fluids (Hartman's solution), as part of routine care. The study intervention (open placebo) is based on injection of placebo into an infusion bag accompanied by the verbal explanation. The placebo is 5 ml NaCl 0.9%.
  Interventions: Behavioral: Open Label Placebo

INTERVENTIONS:
Behavioral: Open Label Placebo — Any woman who arrive to the labor room is connected to fluids (Hartman's solution), as part of routine care. The study intervention (open placebo) is based on injection of placebo into an infusion bag accompanied by a verbal suggustion. The placebo is 5 ml NaCl 0.9%.
  Arms: Open placebo

SUMMARY:
The human nervous system continuously processes a potentially overwhelming stream of signals from bodily senses, which induces uncertainty. To reduce this uncertainty, the brain transforms sensory input into a reliable perception of the world. According to the Bayesian hypothesis of perception, based on probabilistic estimation, conscious perception is shaped by both the current state of sensory information and by past experiences, associative learning, stored memories, and beliefs. This framework is particularly relevant for explaining the phenomenon of pain, including individual differences in pain perception and response.

The focus of the present work is pain during childbirth, representing a major acute pain event. Pain during childbirth is a complex and unique experience with both sensory and emotional components, embedded within a defined physiological process. A key concept of the Bayesian model related to pain perception is the placebo phenomenon, which offers a compelling explanation for the analgesic placebo response.

The overarching aim of this study is to evaluate whether the Bayesian model can account for changes in pain perception during labor following open placebo administration, as well as the involvement of expectations and personality traits.

The study will be conducted at Hillel-Yaffe Medical Center, with the participation of 120 pregnant women. The research will be divided into two stages. The first stage will occur during the prenatal period, while participants are in a pain-free state. During this stage, questionnaires will be completed to assess expectations and personality traits, and the Focused Analgesia Selection Test (FAST) will be administered to evaluate within-subject variability in pain intensity. The second stage will take place during labor and will involve an open placebo intervention, during which pain levels and analgesic consumption will be monitored.

DETAILED DESCRIPTION:
Aims and Hypotheses

Overall Aim:

To assess whether the Bayesian model can explain changes in pain perception during labor following open-placebo administration.

Specific Aims and Hypotheses:

Aim 1: To investigate whether open placebo reduces pain and analgesic consumption during labor.

Hypothesis 1: As most evidence supporting the efficacy of open placebo originates from chronic pain contexts, and given the intensity of labor pain, this hypothesis is bidirectional-open placebo may or may not modulate pain and analgesic consumption during labor at the group level.

Aim 2: To examine whether FAST outcomes predict changes in pain and analgesic consumption during labor following open-placebo administration.

Hypothesis 2: FAST outcomes will predict changes in pain and analgesic use. Lower within-subject variability in pain reports during FAST will be associated with smaller changes in pain and analgesic consumption following open placebo.

Aim 3: To explore the role of expectations and personality traits in placebo analgesia and their potential moderating effects on the relationship between FAST outcomes and the placebo response during labor.

Hypothesis 3.1: Personality traits associated with the prior function will moderate the relationship between FAST outcomes and the placebo response.

Hypothesis 3.2: Personality traits associated with the likelihood function will not moderate this relationship.

Methods

1. Participants:

   Participants will include pregnant women admitted to Hillel Yaffe Medical Center. Based on power analysis (t-test, medium effect size = 0.5, α = 0.05, power = 0.8, allocation ratio = 0.666), a sample size of 106 is required. To compensate for potential dropouts, 120 participants will be recruited.

   Inclusion criteria:

   Singleton pregnancy after 24 weeks of gestation

   No contraindications for analgesia or vaginal birth

   Exclusion criteria:

   Obstetric emergencies such as intrauterine death, suspected placental separation, uterine rupture, placenta previa, or scheduled cesarean section
2. Tools and Procedures 2.1. Pain Assessment Pain will be measured using the Visual Analogue Scale (VAS), a unidimensional tool asking participants to rate pain from 0 ("no pain") to 10 ("worst imaginable pain"). Assessments will occur every 60 minutes throughout labor.

   2.2. Analgesic Consumption Assessment Analgesia at Hillel Yaffe Medical Center includes intravenous Pethidine and epidural anesthesia. Nitrous oxide is not available due to infrastructure limitations. Analgesic usage will be tracked via medical records and epidural pump data, including usage duration, PCA button presses, and administered doses.

   2.3. FAST Assessment The Focused Analgesia Selection Test (FAST) evaluates variability in response to noxious thermal stimuli of varying intensities, applied to the ventral surface of the non-dominant arm using a thermal sensory analyzer. Pain ratings (0-100 scale) are recorded after each stimulus delivered every 20 seconds. Variability is quantified using R² and ICC values. Lower variability indicates higher confidence in sensory input. Test duration is approximately 20 minutes. FAST outcomes are expected to positively correlate with changes in clinical pain.

   2.4. Open Placebo Intervention

   Upon admission to the delivery room, participants receive standard Ringer solution. Participants will be randomly assigned to one of two groups:

   Open Placebo Group: The midwife will explain that although the infusion contains no medication, previous research has shown it may reduce pain.

   Control Group: The standard explanation will be provided, stating the fluids are intended only to maintain venous access.

   Placebo response will be assessed through:

   Differences in pain intensity (area under the curve of VAS scores over time) between groups

   Differences in analgesic consumption, particularly fentanyl dosage via PCA, between groups

   Analyses will also consider placebo response during distinct labor stages.

   2.5. Expectations Assessment

   Expectations will be measured using two questionnaires:

   A short-form expectation questionnaire with items on treatment expectations and hopes.

   A childbirth-specific questionnaire measuring fear and expectations surrounding birth, using a 6-point Likert scale, with higher scores indicating greater fear.

   2.6. Personality Characteristics Assessment

   Suggestibility:

   Measured using the Short Suggestibility Scale (SSS), consisting of 21 items. Higher scores indicate greater suggestibility.

   Anxiety:

   Assessed with the GAD-7, a 7-item scale ranging from 0 to 3 per item, with a total score from 0 to 21. Higher scores reflect more severe anxiety symptoms.

   Interoception:

   Evaluated with the Multidimensional Assessment of Interoceptive Awareness (MAIA), comprising 32 items across eight subscales. Items are rated on a 6-point Likert scale.

   Body Awareness:

   Measured using the Body Awareness Questionnaire, an 18-item scale using a 7-point Likert format. Higher scores indicate increased sensitivity to bodily cues.

   Self-Awareness:

   Evaluated using the short version of the Self-Consciousness Scale-Revised (SCS-R), with 23 items assessing private and public self-awareness on a 4-point scale.
3. Study Design The study will be conducted in the Obstetrics Division at Hillel Yaffe Medical Center. Following ethical and regulatory approval, participant recruitment will begin.

Phase 1:

Conducted prior to labor, when participants are pain-free. Participants will complete demographic, medical, and psychological questionnaires and undergo FAST to measure variability in pain reporting.

Phase 2:

Conducted during labor. Participants will be randomized into control or open placebo groups using a 2:1 allocation ratio (favoring the open placebo group). This ratio supports the analyses in Aims 2 and 3. Randomization will be double-blinded; allocation will be concealed using envelopes and administered by independent personnel not involved in labor care or pain assessments.

Pain intensity will be recorded hourly using VAS. Participation concludes post-delivery, before transfer to the maternity ward.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with one fetus who are after 24th week onwards.
* Without contraindications for analgesia at birth.
* Without contraindications for vaginal birth.

Exclusion Criteria:

* Women in obstetric emergencies, including intrauterine death, suspected placental separation, uterine rupture, placental opening
* Elective cesarean section
* Receiving psychiatric treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity on a 0-10 Numerical Pain Scale (NPS) | Each 60 minutes through the labor process.
  Pain assessment will be performed by using the unidimensional Numerical Pain Scale (NPS) by asking the patient to range the pain, subjectively, from her point of view, from none (0) to a worst imaginable pain (10). Pain intensity will be assessed once in 60 minutes for the duration of the labor. Since each labor duration is difrent, the primary outcome would be the levels of pain during the labor process. Those intensities over time will be compared bewteen the two study arms. In addition, in additional analyses, pain intensities will be compared for each labor phase, seperatly.
Within-subject variability of pain reports | At baseline
  The Focused Analgesia Selection Test (FAST) procedure will be used to assess the within-subject variability of pain reports. The FAST includes exposure to several thermal noxious stimuli, administrated repeatedly at different intensities, which will be delivered to the ventral surface of the non-dominant arm (Medoc® Thermal Sensory Analyzer II with a thermodin size of 30 * 30 mm). Pain intensity ratings are obtained from the participant after each stimulus on a 0-100 numerical rating scale (NRS) ranging from 0 ("no pain") to 100 ("worst pain imaginable"). Stimuli will be triggered automatically every 20 seconds. Relationship between stimulus intensities and pain reports are calculated (R2 and ICC) to assess the magnitude of variability observed.

SECONDARY OUTCOMES:
Assessment of expectations from the treatment | At baseline
  Patients' expectations toward the treatment will be assessed by the EXPECT questionnaire (short version), which includes four items. Three items relate to the respondent's realistic expectations from the treatment, and one item relates to his/her hopes and wishes regarding the treatment. The intent of the question about hope is to increase respondents' focus on answering the 3 expectations questions in terms of their realistic expectations as opposed to their hopes for treatment outcomes. Alpha Cronbach for the short form of the EXPECT questionnaire is 0.89 according to the authors' report.
Fear of childbirth | At baseline
  Severe fear of childbirth will be measured by the Wijma Delivery Expectancy/Experience Questionnaire (W-DEQ), 27 Version A. The W-DEQ consists of 33 items, all of which are rated on a 6-point Likert scale, ranging from 0 to 5. Sum scores range from 0 to 165, with higher scores reflecting a greater degree of fear of childbirth. As suggested in the literature, participants with sum scores ≥85 were defined as suffering from severe fear of childbirth. Internal consistency of the W-DEQ in our study sample was high, with Cronbach's α = .92. The questionnaire has been translated and back-translated by Yael Benyamini and her research team.
Suggestibility | At baseline
  To assess the suggestibility, we are going to use short suggestibility scale (SSS) from the Multidimensional Iowa Suggestibility questionnaire, a scale of multidimensional measure of suggestibility with two companion constructs, with 95 items in total. In the original study by Kotov and colleagues the SSS scale reliability was .89 and correlated with the total suggestibility index obtained with the Multidimensional Iowa Suggestibility Scale. The SSS is composed by 34 21 items, and calculated by the sum of each item, and higher scores represent higher suggestibility trait.
Anxiety | At baseline
  Anxiety will be measured by the Generalized Anxiety Disorder Questionnaire (GAD-7). The GAD-7 is a seven items self-report scale to assess the frequency of symptoms of anxiety with a 4-point Likert-scale ranging from 0 (not at all) to 3 (nearly every day). Items are summed to yield a total score ranging from 0 to 21, with higher scores indicating more anxiety symptoms. The GAD-7 has good sensitivity and specificity for specific anxiety disorders. The GAD- 7 severity cut point is 10 for moderate and severe anxiety. In this study, we used the sum of the GAD-7 as a continuous variable as well as indication for anxiety disorder using the validate cut-off of ≥10. Cronbach's alpha coefficient for the current study was α = 0.92.
Interoception | At baseline
  This personality trait will be measured by Multidimensional Assessment of Interoceptive Awareness (MAIA). Interoceptive sensibility questionnaire aims to distinguish beneficial from maladaptive interoception attention towards one's senses. The Hebrew version of the MAIA questionnaire includes 32 items and is divided into 8 subscales: (1) noticing; (2) not-distracting; (3) not-worrying; (4) attention regulation; (5) emotional awareness; (6) self-regulation; and (7) trusting. All 32 items are answered on a 6-point Likert scale, ranging from 0 ("never") to 5 ("always"). Higher subscale scores indicate higher levels of positive awareness.
Body Awareness | At baseline
  This feature will be measured by Body Awareness Questionnaire. This questionnaire was developed to assess sensitivity to bodily processes and small changes in functioning, the capability to anticipate bodily reactions to internal and environmental changes. It is an 18-item scale rated on a 7-point Likert scale, ranging from 1 ("not true at all about me") to 7 ("very true about me") , and higher mean scores reflect higher sensitivity to somatic cues. Previous studies demonstrated high reliability (Cronbach's alpha = .82), test-retest reliability (r = .80), and evidence for convergent and discriminant validity.
Self-consciousness | At baseline
  The SCS-R (Self-consciousness scale- revised), in its short version, examines the self-awareness of the subject by assessing two key aspects of self-awareness: private and public. Private self-awareness describes awareness of various aspects (emotional or perceptual) of the subject himself, who is the only one who is aware of them. Public self-awareness refers to the subject's awareness of how he or she is perceived by others. The questionnaire contains 23 self-report items on the Likert scale (0-not like me at all and up to 3 very much like me).
Questionnaire for the prediction of the placebo response | At baseline
  A new Questionnaire that we are developing that will be utilized in this study. It includes 32 itmes, ranging from 0 ("never") to 4 ("always).

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: Yes
Will be shared via online link
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication of results
Access Criteria: Everyone